CLINICAL TRIAL: NCT06856317
Title: Use of a Smartphone APP for the Management of Postoperative Home Recovery: an Exploratory Study
Brief Title: Use of a Smartphone APP for the Management of Postoperative Home Recovery
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: APPCHTOR
Record Dates: First submitted 2025-01-10; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-12

CONDITIONS: Rehospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To calculate the incidence rates of postoperative adverse events (moderate and severe) and rehospitalization in patients undergoing thoracic surgery followed in follow-up using a smartphone application.

DETAILED DESCRIPTION:
This is an observational, exploratory, cohort, retrospective study. For this study, data acquired on patients who participated in the trial period of the app will be retrospectively analyzed. Our Operating Unit used the care4today app on a trial basis during the period between March 1 and October 31, 2023, focusing on monitoring the first 30 days after discharge. The app was offered to patients scheduled for thoracic surgery involving access to the pleura. After a few setup questions, the app was activated upon discharge. For the first 15 days it sent daily questions via notification regarding general health status, postoperative pain, respiratory capacity, and resumption of activities. From day 15 to day 30 after discharge, questions were asked every 4 days. All relevant responses were forwarded via e-mail to the clinician in the form of an orange or red alert in relation to lesser or greater severity.

Patients were treated according to clinical practice in accordance with the clinician's judgment and the information in the Data Sheet of each individual product of any concomitant therapies administered according to clinical practice. Informed consent will be collected during follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patients undergoing thoracic surgery
* Patients who used the care4today app
* Obtaining informed consent to participate in the study

Exclusion Criteria:

* nothing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the study, the researchers expect to enroll the 96 patients who participated in the trial period of the application.
  Considering the 30-day incidence and re-hospitalization rates as sample proportions of 0.5 (most conservative assumption), a numerosity of 96 will be sufficient to estimate the proportions with bilateral 95% confidence intervals of 0.2.
  The width of the confidence interval was calculated using PASS 2023, version 23.0.2.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Adverse event rate | 30 days after surgery
  Complications are reported by patients using the mobile phone app.
Moderate adverse event rate | 30 days after surgery
  Complications are reported by patients using the mobile phone app.
Severe adverse event rate | 30 days after surgery
  Complications are reported by patients using the mobile phone app.
Rehospitalization rate | At 30 days from surgery
  Rehospitalization rate in the first 30 days from home discharge.

SECONDARY OUTCOMES:
Non-response rate to questions asked by the application | Throughout the study period, an average of 30 days
  Use of the app

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Bertoglio, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero Universitaria di Bologna, Bologna, Emilia-Romagna, Italy